CLINICAL TRIAL: NCT00059514
Title: Arab American Youth: Tobacco Use and Intervention
Brief Title: Tobacco Use Among Arab American Youth
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Virginia H. Rice, Principal Investigator, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Organization: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: 5R01HD37498-3; 5R01HD037498 (NIH)
Record Dates: First submitted 2003-04-28; First posted 2003-04-29 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Tobacco Use Disorder
Keywords: Youth; Adolescents; Smoking cessation; Smoking prevention; Risk factors; Arab Americans
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Modified Project Toward No Tobacco Use

SUMMARY:
Michigan has the 10th highest smoking rate in the nation. Smoking rates are also very high in the Middle East and in Arab American families. The purpose of this study is to learn about tobacco use in Michigan Arab American youth ages 14 to 18. The study will evaluate why some young people start smoking and others do not. The study will also test an educational program designed to encourage young people to either quit tobacco use or to avoid it.

DETAILED DESCRIPTION:
Cigarette smoking is the chief avoidable cause of death and disease in Michigan, the United States, and the world. In 1996, 25.9% of the Michigan adult population smoked cigarettes; Michigan has the 10th highest smoking rate in the nation. When the indirect costs of lost income due to smoking-related illnesses and premature death are added to the cost of medical care, tobacco use costs Michigan citizens more than $2.6 billion per year (Michigan Department of Community Health (MDCH), 1996). Contributing to tobacco use statistics in Michigan is a rapidly growing Arab American immigrant population. Studies have shown cigarette smoking rates in Middle-Eastern adolescents range from 33% to 58%. This study will examine cultural, personal, social, and environmental forces operating in Arab American youths at risk for habitual tobacco use. The study will also test the effects of a smoking cessation/prevention intervention on smoking behavior.

The settings for this study are the Arab Community Center for Economic and Social Services (ACCESS) Teen Health Center, which services almost 2,500 youth visits each year, and local high schools with a significant population of Arab American youth. The majority of the people served by the clinic are poor, under-educated, live in extended families of 3 to 5 adults, are immigrants, and speak Arabic as a first language. A total of 4,000 adolescents over 14 years old will be asked to provide information on demographic and cultural variables, self-esteem, stress, family and peer tobacco use, intention to use tobacco, history of tobacco use, initial stage of change, and perceived health.

Youths with the highest risk for tobacco use will be randomly assigned to either a Modified Project Toward No Tobacco Use (Project TNT) intervention or a wait list control group. Project TNT, the precursor to the Arab American-specific modified Project TNT, was designed to target the primary causes of tobacco use among adolescents and has been shown to be effective in diverse cultural groups. The modified Project TNT consists of weekly 40-minute sessions with a health educator over 4 weeks. Bilingual health educators will deliver the intervention in a small group (four to six adolescents) or classroom context. Follow-up data will be collected at 3, 6, and 12 months after the program is completed. Youth assigned to the wait list control group will participate in the modified Project TNT after the Month 6 follow-up data is collected from the first group.

ELIGIBILITY:
Inclusion Criteria

* 14-18 years
* Self-identify as Arab American
* Attendee of a teen health clinic or high school

Exclusion Criteria

* older than 18 years
* does not identify as Arab or Arab American

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 2300 + school-based Arab American adolescents (14-18 years) were recruited for participation in this study of tobacco use.
  1700 students provided detailed health and tobacco use histories. 616 students were assigned by classroom to a smoking cessation intervention or to a class on health.
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Actual)
Dates: Start 2000-05 (Actual); Primary Completion 2005-04 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia H Rice, PhD, RN, Principal Investigator — Wayne State University
Locations (1):
- Arab American Center for Economic & Social Services, Dearborn, Michigan, United States

IPD SHARING:
Plan to Share IPD: No